CLINICAL TRIAL: NCT05106894
Title: Mobile Health Intervention to Promote Positive Infant Health Outcomes in Guatemala
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Children's Hospital Los Angeles (Other)
Collaborators: Wuqu' Kawoq, Maya Health Alliance (Other); Eunice Kennedy Shriver National Institute of Child Health and Human Development (NICHD) (NIH)
Responsible Party: Principal Investigator, Beth Smith, Principal Investigator, Children's Hospital Los Angeles
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: CHLA-21-00168; 5R21HD107983 (NIH)
Record Dates: First submitted 2021-10-25; First posted 2021-11-04 (Actual); Results first posted 2025-05-28 (Actual); Last update posted 2025-05-28 (Actual); Status verified 2025-05

CONDITIONS: Infant Development

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- smartphone application to promote nurturing care (Experimental): a caregiver-directed smartphone application will directly engage first-time caregivers in providing nurturing care
  Interventions: Behavioral: smartphone application to promote nurturing care
- printed caregiving materials (Active Comparator): caregivers will receive print materials on early childhood stimulation
  Interventions: Behavioral: printed caregiving materials

INTERVENTIONS:
Behavioral: smartphone application to promote nurturing care — see arm description
  Arms: smartphone application to promote nurturing care
Behavioral: printed caregiving materials — see arm description
  Arms: printed caregiving materials

SUMMARY:
Promoting optimal development for children at risk in low- and middle-income countries (LMICs) is an important global health priority. Supporting caregivers to provide nurturing care is an evidence-based strategy, however feasibility of scaling-up this supporting is limited by competing demands on health workers' time. For infant development, mHealth technologies have the potential to solve this problem by providing tailored content directly to caregivers, involving and empowering them to promote infant development, promoting and facilitating interactions with health workers when areas of concern are identified and, therefore, expanding the reach of healthcare systems. This overall study is designed to explore this idea, by designing a caregiver-directed smartphone application to directly engage first-time caregivers in rural Guatemala in providing nurturing care and, after design, to conduct a prospective implementation trial of its use followed by an adequately-powered efficacy study.

DETAILED DESCRIPTION:
Rationale: According to recent estimates, 43% of children under age 5 residing in low- and middle-income countries (LMICs)-250 million children in total-are at risk of not reaching their developmental potential due to living in environments with malnutrition, poverty, and lack of early stimulation. Mobile health (mHealth) technology represents an efficient strategy for scaling interventions to promote infant development.

Intervention: Pilot randomized controlled trial of mHealth application compared to paper caregiving materials. Length of intervention = 6 months.

Objectives and purpose: We will test a smartphone application that will directly engage caregivers in providing nurturing care to at-risk infants. We will assess effectiveness of the mHealth application compared to paper caregiving materials by establishing effect sizes of group differences in Bayley scores after 6 months.

Study population: newborn infants.

ELIGIBILITY:
Inclusion Criteria:

* first-time caregivers with an infant in the eligible age range (0-4 weeks)
* infant from singleton birth
* infant from full-term (> 37 weeks gestation) birth

Exclusion Criteria:

* Presence of acute malnutrition/wasting or severe medical illness (heart disease, kidney disease, congenital abnormality) in the infant
* medical need for supplementation of breastfeeding
* caregiver not literate

Max Age: 6 Months | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 41 (Actual)
Dates: Start 2023-01-11 (Actual); Primary Completion 2024-08-31 (Actual); Study Completion 2024-08-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Beth A Smith, PT, DPT, PhD, Principal Investigator — Children's Hospital Los Angeles
Locations (1):
- Wuqu' Kawoq/ Maya Health Alliance, Chimaltenango, Guatemala

IPD SHARING:
Plan to Share IPD: Yes
de-identified data will be shared via NICHD DASH
Supporting Information: Study Protocol
Time Frame: data will become available upon completion of the study and will remain available indefinitely.

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were recruited from January 2023 to March 2023.
Pre-assignment Details: Participants were infants. The Enrollment number and number of participants Started/Completed represents individual infants.
Period: Overall Study
Arm/Group | Smartphone Application to Promote Nurturing Care | Printed Caregiving Materials
Started | 20 | 21
Completed | 19 | 21
Not Completed | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Smartphone Application to Promote Nurturing Care | Printed Caregiving Materials | Total
Number analyzed (Participants) | 19 | 21 | 40
Age, Continuous [Median (Inter-Quartile Range); unit: days] | 20 [13 to 24] | 14 [9 to 16] | 17 [11 to 20]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 10 | 13 | 23
  Male | 9 | 8 | 17
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Maya ethnicity | 18 | 20 | 38
Region of Enrollment [Number; unit: participants]
  Guatemala | 19 | 21 | 40

OUTCOME MEASURES:

1. Primary Outcome: Bayley Composite Scores After 6 Months, Effect Size of Group Difference: COGNITIVE
Description: Bayley Scales of Infant and Toddler Development (4th edition). Composite scores are norm-referenced based on age. Higher scores are better. Minimum composite score value is 60 and maximum composite score value is 140.
Time Frame: 6 months
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Smartphone Application to Promote Nurturing Care | Printed Caregiving Materials
Number analyzed (Participants) | 19 | 20
score on a scale | 111 (9) | 111 (10)
Statistical Analysis 1: Comparison: Smartphone Application to Promote Nurturing Care vs Printed Caregiving Materials; Test type: Equivalence — Adjusted difference between groups in composite scores calculated using an ordinary least squares linear regression model (with adjustments for sex of child, caregiver educational level, poverty score, birth weight and change in length for age Z score from 0 to 6 months); Median Difference (Final Values) = -1.0, 95% CI 2-sided [-7.4 to 5.5]

2. Primary Outcome: Bayley Composite Scores After 6 Months, Effect Size of Group Difference: MOTOR
Description: as for outcome 1
Time Frame: 6 months
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Smartphone Application to Promote Nurturing Care | Printed Caregiving Materials
Number analyzed (Participants) | 19 | 20
score on a scale | 105 (9) | 106 (11)
Statistical Analysis 1: Comparison: Smartphone Application to Promote Nurturing Care vs Printed Caregiving Materials; Test type: Equivalence — [test comment as in outcome 1, analysis 1]; Median Difference (Final Values) = -2.3, 95% CI 2-sided [-8.3 to 3.6]

3. Primary Outcome: Bayley Composite Scores After 6 Months, Effect Size of Group Difference: LANGUAGE
Description: as for outcome 1
Time Frame: 6 months
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Smartphone Application to Promote Nurturing Care | Printed Caregiving Materials
Number analyzed (Participants) | 19 | 20
score on a scale | 104 (6) | 104 (6)
Statistical Analysis 1: Comparison: Smartphone Application to Promote Nurturing Care vs Printed Caregiving Materials; Test type: Equivalence — [test comment as in outcome 1, analysis 1]; Mean Difference (Final Values) = -1.8, 95% CI 2-sided [-5.6 to 2.1]

ADVERSE EVENTS:
Time Frame: 6 months
Description: The IRB's determined that the research involves no greater than minimal risk. Data were monitored on an ongoing basis by the PI.
Arm/Group | Smartphone Application to Promote Nurturing Care | Printed Caregiving Materials
All-Cause Mortality (participants affected / at risk) | 0/19 | 0/21
Serious Adverse Events (participants affected / at risk) | 0/19 | 0/21
Other Adverse Events (participants affected / at risk) | 0/19 | 0/21

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2023-08-09): https://cdn.clinicaltrials.gov/large-docs/94/NCT05106894/Prot_SAP_000.pdf
  • Informed Consent Form (2022-10-26): https://cdn.clinicaltrials.gov/large-docs/94/NCT05106894/ICF_001.pdf